CLINICAL TRIAL: NCT02510183
Title: Evaluation of the Effects of P6 Acupressure Application on Postoperative Nausea and Vomiting Before Laparoscopic Cholecystectomy
Brief Title: P6 Acupressure Before Laparoscopic Cholecystectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: GulhaneMMA
Record Dates: First submitted 2015-06-28; First posted 2015-07-29 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-06

CONDITIONS: Postoperative Complications; Postoperative Nausea and Vomiting
Keywords: Acupressure; Perioperative Care; Postoperative Nausea and Vomiting; Nursing Care Management
MeSH Terms: conditions — Postoperative Complications; Postoperative Nausea and Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acupressure Wrist Band (Active Comparator): Patient receive preoperative education a day before surgery, education for acupressure application on the day of surgery, an acupressure wrist band is applied on P6 acupoint in both wrist an hour before surgery
  Interventions: Device: Acupressure Wrist Band
- Placebo Wrist Band (Placebo Comparator): Patient receive preoperative education a day before surgery, an placebo acupressure wrist band is applied in both wrist an hour before surgery
  Interventions: Device: Placebo Acupressure Wrist Band
- Control Grup Without Band (No Intervention): Patient receive preoperative education a day before surgery, and patient are only visited an hour before surgery

INTERVENTIONS:
Device: Acupressure Wrist Band — Acupressure wrist band is a knitted elasticated wrist band, which operates by applying pressure on the P6 acupressure point on each wrist by means of a plastic stud.
  Other Names: Sea Band
  Arms: Acupressure Wrist Band
Device: Placebo Acupressure Wrist Band — Placebo Acupressure Wrist Band is a knitted elasticated wrist band without a plastic stud.
  Arms: Placebo Wrist Band

SUMMARY:
This study is to evaluate the effect of preoperative acupressure application on Postoperative nausea and vomiting (PONV) in patients undergoing laparoscopic cholecystectomy in terms of being in high risk group for PONV.

DETAILED DESCRIPTION:
Prevention of postoperative complications is one of the main tasks of nurses. However, there are limited nursing interventions that can be done to prevent PONV. The American Society of PeriAnesthesia Nurses suggest nurses to teach patients with a high risk of PONV about acupressure application on P6 acupoint or to apply acupressure wristbands preoperatively. However this suggestion has a low evidence.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing elective laparoscopic cholecystectomy
* Patients who make their admission the day before surgery
* Patients with American Society of Anesthesiologists (ASA) physical status classification system I and II
* Patient who gave written consent to participate in the study

Exclusion Criteria:

* Patient who undergone urgent laparoscopic cholecystectomy
* Patients who make their admission on the day of surgery
* Patients with who do not conform physical status of ASA I and II
* Patients who loss single or both upper extremity
* Patients with open wounds, scar tissue or infection on wrist in acupressure application area

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2015-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Acupressure affect on Postoperative Nausea, Vomiting and medication need | 24 hours postoperatively
  Postoperative nausea, vomiting and medication need are assessed on 2nd, 6th and 24th hours postoperative. Nausea severity measured by 0-10 scoring (0- no nausea,10- nausea as bad as can be), and vomiting is assessed as episodes. Number of antiemetics and analgesics medications that are given (out of routine therapy) are also evaluated.

SECONDARY OUTCOMES:
Pain | 24 hours postoperatively
  Pain measured by 0-10 scoring (0- no pain,10- pain as bad as can be) on 2nd, 6th and 24th hours postoperative.
Perioperative Stress | 48 hour
  Perioperative Stress measured by State-Trait Anxiety Inventory (STAI) score on day before surgery and day after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Emine Iyigun, Assoc.Prof., Study Chair — Gulhane Military Medical Academy, School of Nursing, Department of Surgical Nursing; Mehmet F CAN, Assoc.Prof., Study Chair — Gulhane Military Medical Academy, Department of General Surgery; Sibel Yilmaz Sahin, PhDs, Principal Investigator — Gulhane Military Medical Academy, School of Nursing, Department of Surgical Nursing

REFERENCES:
- [Background] Adib-Hajbaghery M, Etri M, Hosseainian M, Mousavi MS. Pressure to the p6 acupoint and post-appendectomy pain, nausea, and vomiting: a randomized clinical trial. J Caring Sci. 2013 Jun 1;2(2):115-22. doi: 10.5681/jcs.2013.014. eCollection 2013 Jun. PMID 25276717
- [Background] Agarwal A, Bose N, Gaur A, Singh U, Gupta MK, Singh D. Acupressure and ondansetron for postoperative nausea and vomiting after laparoscopic cholecystectomy. Can J Anaesth. 2002 Jun-Jul;49(6):554-60. doi: 10.1007/BF03017380. PMID 12067865
- [Background] American Society of PeriAnesthesia Nurses PONV/PDNV Strategic Work Team. ASPAN'S evidence-based clinical practice guideline for the prevention and/or management of PONV/PDNV. J Perianesth Nurs. 2006 Aug;21(4):230-50. doi: 10.1016/j.jopan.2006.06.003. No abstract available. PMID 16935735
- [Background] Hickman AG, Bell DM, Preston JC. Acupressure and postoperative nausea and vomiting. AANA J. 2005 Oct;73(5):379-85. PMID 16261854
- [Background] Lee A, Fan LT. Stimulation of the wrist acupuncture point P6 for preventing postoperative nausea and vomiting. Cochrane Database Syst Rev. 2009 Apr 15;(2):CD003281. doi: 10.1002/14651858.CD003281.pub3. PMID 19370583
- [Background] Sadati L, Pazouki A, Mehdizadeh A, Shoar S, Tamannaie Z, Chaichian S. Effect of preoperative nursing visit on preoperative anxiety and postoperative complications in candidates for laparoscopic cholecystectomy: a randomized clinical trial. Scand J Caring Sci. 2013 Dec;27(4):994-8. doi: 10.1111/scs.12022. Epub 2013 Jan 28. PMID 23350886